CLINICAL TRIAL: NCT04345380
Title: Rotational Stability of the Acrysof, Tecnis and Envista Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Univ. Prof. Dr. med.univ. Rupert Menapace, Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1746/2014
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Cataract; Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

ARMS (3):
- Acrysof Rotation (Active Comparator): Implantation of the Acrysof SN60WF Intraocular lens to the 0 ±10, 45± 10, 90±10 or 135± axis.
  Interventions: Other: Implantation of an Alcon Acrysof SN60WF intraocular lens
- Tecnis Rotation (Active Comparator): Implantation of the Tecnis ZCB00 Intraocular lens to the 0 ±10, 45± 10, 90±10 or 135± axis.
  Interventions: Other: Implantation of an AMO Tecnis ZCB00 intraocular lens
- Envista Rotation (Active Comparator): Implantation of the Envista MX60 Intraocular lens to the 0 ±10, 45± 10, 90±10 or 135± axis.
  Interventions: Other: Implantation of an Envista MX60 intraocular lens

INTERVENTIONS:
Other: Implantation of an Alcon Acrysof SN60WF intraocular lens — Patients suffering from senile cataract getting replaced their human crystalline cataractous lens
  Arms: Acrysof Rotation
Other: Implantation of an AMO Tecnis ZCB00 intraocular lens — Patients suffering from senile cataract getting replaced their human crystalline cataractous lens
  Arms: Tecnis Rotation
Other: Implantation of an Envista MX60 intraocular lens — Patients suffering from senile cataract getting replaced their human crystalline cataractous lens
  Arms: Envista Rotation

SUMMARY:
Brief Summary:

Age-related cataract is the main cause of impaired vision in the elderly population worldwide. In the UK, more than half of people who are over 65 years old have some cataract development in one or both eyes. The only treatment that can restore functional visual ability is cataract surgery where the opacified crystalline lens is removed by phacoemulsification and an artificial intraocular lens is implanted. It is estimated that around 10 million cataract operations are performed around the world each year. Cataract operations are generally very successful, with a low risk of serious complications.

During the past two decades, cataract surgery underwent tremendous change and modernisation resulting in today's small incision phacoemulsification surgery and a safe technique with a short rehabilitation time for the patient. Traditional spherical monofocal intraocular lenses (IOLs) restore best-corrected vision and may lessen the need for spectacles. These IOLs correct only the spherical portion of the total refractive error and do not correct corneal astigmatism. Astigmatism is a visually disabling refractive error affecting the general population, especially those with cataract. At least 15% to 20% of cataract patients have 1.5 diopters (D) or more of corneal or refractive astigmatism. With increased patient expectations, the trend is not only to remove the cataract but also to address the problem of pre-existing astigmatism at the time of surgery.

Surgical-induced astigmatism can be reduced by smaller incisions, i.e. microincision cataract surgery (MICS), which by definition is surgery performed through incisions smaller than 2.0 mm, reducing the need for suturing. This results in better corneal optical quality, thus improving visual outcomes. There are also other surgical options to correct preexisting astigmatism during cataract surgery like: selectively positioning of the phacoemulsification incision; astigmatic keratotomy with corneal or limbal relaxing incisions; excimer laser refractive procedures such as photorefractive keratectomy, laser in situ keratomileusis, and laser-assisted subepithelial keratectomy; or implanting pseudophakic toric posterior chamber intraocular lenses (IOLs).

Toric IOLs have been shown to result in good visual and refractive outcomes. Combined with MICS, these IOLs can allow effective correction of cylindrical errors intraoperatively, improving visual quality and thus leading to spectacle independence. Plate haptic and loop haptic toric IOLs have been considered for about a decade but have been associated with postoperative rotational instability. Rotation of a toric lens from its intended orientation degrades its corrective power, with approximately 3.3% loss of cylindrical power for every degree off axis. A misorientation of approximately 30° negates the effectiveness of astigmatic correction, and a misorientation of more than 30° may induce additional astigmatism. Although some patients are asymptomatic despite induced astigmatism, others experience symptoms such as blurred or distorted vision, headache, fatigue, eyestrain, squinting, or eye discomfort. Thus, IOL orientation stability is an essential goal in toric IOL design.

RATIONALE

The purpose of this study is to assess and compare the axial IOL rotation and optical quality (refraction, visual acuity, decentration and tilt) and capsular bag reaction after micro-incision surgery with an IOL implantation in cataract patients - Acrysof SN60WF, Tecnis ZCB00 & Envista MX60 IOL

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral age-related cataract necessitating phacoemulsification extraction and posterior IOL implantation
* Need for spherical IOL correction between 10.00 and 30.00 D
* Pupil dilation of ≥ 6.5 mm
* Age 40 and older

Exclusion Criteria:

* Corneal abnormality
* Pseudoexfoliation
* Preceding ocular surgery or trauma
* Uncontrolled glaucoma
* Proliferative diabetic retinopathy
* Iris neovascularization
* History of uveitis/iritis
* Microphthalmus
* Recurrent intraocular inflammation of unknown etiology
* Blind fellow eye
* Uncontrolled systemic or ocular disease
* Pregnancy and lactation

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Rotational stability from End of Surgery to 6 months | 4-7 months
  Change in axis position of an intraocular lens Alcon SN60WF, AMO Tecnis ZCB00 or Bausch&Lomb Envista MX60 from end of surgery (baseline axis) to 1 hour, 1 week, 1 month and 4-7 months (end of study visit). The change in axis position will be evaluated with respect to the baseline measurement at the end of surgery. Differences in axis position will be described as rotation in degrees (0 to 360°)

SECONDARY OUTCOMES:
Decentration | 4 to 7 months
  Decentration of the intraocular lens Alcon SN60WF, AMO Tecnis ZCB00 or Bausch&Lomb Envista MX60 will be measured with a Purkinje Meter. Decentration will be described as "Decentration in milimeter"
Tilt | 4 to 7 months
  Tilt of the intraocular lens Alcon SN60WF, AMO Tecnis ZCB00 or Bausch&Lomb Envista MX60 will be measured with a Purkionje Meter. Tilt will be described as "Tilt in degrees at a certain axis"

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna Allgemeines Krankenhaus, Vienna, Austria